CLINICAL TRIAL: NCT00000393
Title: A Phase I Trial of Peptide T: Efficacy for the Neuropsychiatric Complications of Acquired Immunodeficiency Syndrome (AIDS).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 89 MH-28
Record Dates: First submitted 2000-01-17; First posted 2000-01-18 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2002-04

CONDITIONS: HIV Infections; Cognition Disorders
Keywords: Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Cognition Disorders; Acquired Immunodeficiency Syndrome | interventions — Peptide T

INTERVENTIONS:
Drug: Peptide T

SUMMARY:
To study the safety, toxicology, and activity of Peptide T (D-Ala-1-peptide-T-amide) in humans and to find out more about the ability of peptide T to prevent, halt, and/or reverse AIDS-associated immunologic disturbances.

Recent information suggests that the central nervous system (CNS) is often impaired in HIV-infected individuals. The dysfunction of the CNS may be either a direct or an indirect result of HIV infection. One method to prevent HIV infection is to block entry of the virus into the cells of the body. Peptide T shows laboratory evidence of blocking the entrance of HIV into cells that are susceptible to HIV infection. Studies that have been done indicate that peptide T is nontoxic in the doses that are used in this study.

AIDS patients with minimal (group 1) or moderate (group 2) cognitive dysfunction (mental impairment) receive an increasing schedule of three dosage levels of peptide T. All patients receive an intravenous (IV) dose of peptide T for 10 days followed by the intermediate dose and then the highest dose, each intravenously for 10 days. Following successful completion of 3 IV doses, four patients participate in an intranasal pharmacokinetic (blood level study) dosage trial of 3 doses (different from IV) of peptide T once for each of 3 successive days. Follow-up continues for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* History of either opportunistic infection and/or Kaposi's sarcoma, and/or serologic evidence of past infection with HIV. Ability to give informed consent.
* Allowed but discouraged: Antiretroviral medication. Immunomodulating medication. Psychoactive medication.
* Not breast-feeding
* Abstinence or agree to use barrier methods of birth control / contraception during the study
* Not pregnant
* Negative pregnancy test
* CD4 >= 200 cells/mm3 (200 - 300 - 400 - 500 - 600 - 700 - 800 plus).
* Creatinine <= 1.6 mg/dl
* Hemoglobin >= 12 g/dl
* Platelet Count >= 100000 /mm3

Exclusion Criteria:

* Patients with the following diseases or symptoms are excluded: Space-occupying lesion in brain. Life-threatening opportunistic infection at time of entry into trial. History of major psychiatric illness prior to 1977 or time of initial exposure to HIV, if that is known.
* Patients with the following diseases or symptoms are excluded: Space-occupying lesion in brain. Life-threatening opportunistic infection at time of entry into trial. History of major psychiatric illness prior to 1977 or time of initial exposure to HIV, if that is known.
* Excluded within 4 weeks of study entry:

Antiretroviral agents. Anticancer treatments. Psychoactive agents.

Excluded within 4 months of study entry:

Suramin.

* Avoid: Antiretroviral medication. Immunomodulating medication. Psychoactive medication.
* Excluded within 4 weeks of study entry:

Radiation.

* Breast-feeding
* Positive pregnancy test
* Pregnant
* No abstinence or no agreement to use barrier methods of birth control / contraception during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 1988-01; Primary Completion 1990-01 (Actual)

PRIMARY OUTCOMES:
Patients performance on neuropsychological tests | 10 days plus 10 days plus 3 days
  The additional 3 days was for only 4 patients with follow-up for 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bridge TP, Study Chair — National Institute of Mental Health (NIMH)
Locations (1):
- Los Angeles County - USC Med Ctr, Los Angeles, California, United States